CLINICAL TRIAL: NCT03840122
Title: Comparing ACB + IPACK Block With or Without Local Infiltration in Patients Undergoing Primary Robotic Arm-Assisted TKA
Brief Title: ACB + IPACK Block With or Without Local Infiltration in RA-TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The P.I. decided to cancel this study. On 10/08/19, a study closure request was submitted to the IRB.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Professor, Adult Reconstruction, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18.1246
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Knee Arthropathy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - ACB + IPACK with injection (Experimental): 50 arms: ACB + IPACK block with injection of local anesthetic of Ropivacaine, Epinephrine, Ketorolac, Clonidine and saline
  Interventions: Other: ACB + IPACK block with injection of local anesthetic
- B - ACB + IPACK without injection (Active Comparator): 50 arms: ACB + IPACK block without injection of local anesthetic
  Interventions: Other: ACB + IPACK block without injection

INTERVENTIONS:
Other: ACB + IPACK block with injection of local anesthetic — ACB + IPACK block with injection of local anesthetic which is comprised of the following agents and amounts:
  * Ropivacaine 5mg/ml (49.25ml)
  * Epinephrine 1mg/ml (0.5ml)
  * Ketorolac 30mg/ml (1ml)
  * Clonidine 0.1mg/ml (0.8ml)
  * Saline 48.45ml
  Arms: A - ACB + IPACK with injection
Other: ACB + IPACK block without injection — ACB + IPACK block without an injection of local anesthetic
  Arms: B - ACB + IPACK without injection

SUMMARY:
The purpose of this study is to compare the outcomes of an Adductor canal block (ACB) + interspace between the popliteal artery and the capsule of the knee (IPACK) block along with a single intraoperative injection of a standard local anesthetic that includes Ropivacaine, Epinephrine, Ketorolac, Clonidine and saline to an ACB + IPACK block without the intraoperative injection of a standard local anesthetic in patients undergoing Robotic Arm-Assisted TKA (RA-TKA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over the age of 21
2. Patient is scheduled to undergo a unilateral, primary TKA, secondary to osteoarthritis
3. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization documents
4. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 21
2. Patient's primary diagnosis is not osteoarthritis (e.g. post-traumatic arthritis)
3. Patient is scheduled to undergo a bilateral TKA surgery
4. Patient is unable to read and speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
total length of hospital stay | outcome measure will be taken at 2 weeks postoperatively
  total length of hospital stay as defined by number of days from date of surgery to date of discharge
Knee Society Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery) and 6 weeks (± 2 weeks) postoperatively.
  Knee Society Score as recorded preoperatively and 6 weeks (± 2 weeks) postoperatively. The score is on a scale from 0-100. A higher value represents a better outcome.
WOMAC score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery) and 6 weeks (± 2 weeks) postoperatively
  WOMAC score as recorded preoperatively and 6 weeks (± 2 weeks) postoperatively. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome.
Visual Analog Scale | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively.
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Amount of narcotic medication utilized | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Ability to rise from a chair independently | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Ability to rise from a chair independently (Yes/No)
Active range-of-motion (ROM) | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Distance that patient is able to walk | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Distance that patient is able to walk, as measured in feet
Use of an ambulatory assistive device | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, 6 weeks (± 2 weeks) postoperatively
  Use of an ambulatory assistive device (Yes/No)
Return to driving | outcome measure will be taken 2 weeks (± 4 days) postoperatively and 6 weeks (± 2 weeks) postoperatively
  Return to driving (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Malkani, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No